CLINICAL TRIAL: NCT00623129
Title: Electroacupuncture for Xerostomia in Head and Neck Patients
Brief Title: Electroacupuncture in Treating Chronic Dry Mouth Caused By Radiation Therapy in Patients With Head and Neck Cancer
Status: Terminated | Phase: Not Applicable | Type: Interventional
Why Stopped: Slow accrual; did not meet accrual goal
Sponsor: Mayo Clinic (Other)
Collaborators: National Cancer Institute (NCI) (NIH)
Responsible Party: Sponsor
Allocation: Randomized | Masking: Single | Purpose: Supportive Care
Other Study IDs: CDR0000583031; P30CA015083 (NIH); MCS285 (Other: Mayo Clinic IRB); 2327-05 (Other: Mayo Clinic IRB); NCI-2010-01835 (Registry Identifier: NCI-CTRO)
Record Dates: First submitted 2008-02-22; First posted 2008-02-25 (Estimated); Last update posted 2016-04-19 (Estimated); Status verified 2011-08

CONDITIONS: Head and Neck Cancer; Radiation Toxicity; Xerostomia
Keywords: hypopharyngeal cancer; lip and oral cavity cancer; laryngeal cancer; nasopharyngeal cancer; oropharyngeal cancer; paranasal sinus and nasal cavity cancer; salivary gland cancer; xerostomia; radiation toxicity
MeSH Terms: conditions — Head and Neck Neoplasms; Radiation Injuries; Xerostomia; Hypopharyngeal Neoplasms; Mouth Neoplasms; Laryngeal Neoplasms; Nasopharyngeal Neoplasms; Oropharyngeal Neoplasms; Salivary Gland Neoplasms | interventions — Electroacupuncture

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

INTERVENTIONS:
Other: questionnaire administration
Procedure: electroacupuncture therapy
Procedure: management of therapy complications
Procedure: quality-of-life assessment

SUMMARY:
RATIONALE: Electroacupuncture may help relieve chronic dry mouth caused by radiation therapy. It is not yet known whether electroacupuncture is more effective than a placebo in treating chronic dry mouth caused by radiation therapy in patients with head and neck cancer.

PURPOSE: This randomized clinical trial is studying electroacupuncture to see how well it works compared with a placebo in treating chronic dry mouth caused by radiation therapy in patients with head and neck cancer.

DETAILED DESCRIPTION:
OBJECTIVES:

* To determine if electrostimulation using the Liss stimulator can objectively improve salivary flow as measured by sialometry compared to a placebo device in patients with chronic radiation-induced xerostomia and head and neck cancer.
* To determine if electrostimulation using the Liss Stimulator can improve the subjective sensation of mouth dryness compared to a placebo device.
* To characterize the effect of electrostimulation using the Liss stimulator on quality of life compared to a placebo device.

OUTLINE: Patients are randomized to 1 of 2 treatment arms.

* Arm I: Patients undergo placement of electrodes to the following acupuncture points: stomach, liver, pericardium, small intestine, and large intestine. Patients then undergo electro-stimulation of the acupuncture points using the Liss Stimulator for 20 minutes once a day for 10 days and then 3 times a week for 2 weeks.
* Arm II (placebo): Patients undergo placement of electrodes to the following acupuncture points: stomach, liver, pericardium, small intestine, and large intestine. A device that does not produce an electric current is placed over the electrodes for 20 minutes once a day for 10 days and then 3 times a week for 2 weeks.

Patients complete questionnaires, including the Brief Pain Inventory, the Xerostomia Inventory, and a subscale of the University of Washington Head and Neck Symptom Scale, at baseline, on days 5 and 10 of treatment, and at 1, 3, and 6 months after completion of treatment. Sialometry (unstimulated and stimulated whole saliva measurement) is also performed at the same time points.

After completion of study treatment, patients are followed at 1, 3, and 6 months.

ELIGIBILITY:
DISEASE CHARACTERISTICS:

* Diagnosis of primary head and neck cancer
* Has undergone radiotherapy either as primary or adjuvant therapy ≥ 6 months ago

  * One or more parotid glands must have been in the prior radiotherapy field
* Residual xerostomia after radiotherapy deemed to be significant by patient

  * Failed to respond to a trial of pilocarpine for relief of xerostomia

PATIENT CHARACTERISTICS:

* ECOG performance status 0-3
* Life expectancy ≥ 1 year (based on physician's judgment)
* Able to attend the scheduled study treatments
* Alert and mentally competent
* Not pregnant
* Willing to use contraception during study treatment, if of childbearing age
* No history of Sjögren's disease
* No cardiac pacemaker or any other electrical devices permanently implanted within the body (e.g., dorsal column stimulator)

PRIOR CONCURRENT THERAPY:

* See Disease Characteristics
* More than 2 weeks since prior medication that may cause mouth dryness (e.g., antihistamines, narcotics, tricyclic antidepressants)

Ages: 21 Years to 89 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 30 (Estimated)
Dates: Start 2006-02; Primary Completion 2010-11 (Actual)

PRIMARY OUTCOMES:
Salivary flow as measured by sialometry at baseline, on days 5 and 10 of treatment, and at 1, 3, and 6 months after completion of treatment
Subjective sensation of mouth dryness as measured by quality of life questionnaires at baseline, on days 5 and 10 of treatment, and at 1, 3, and 6 months after completion of treatment
Quality of life as measured by quality of life questionnaires at baseline, on days 5 and 10 of treatment, and at 1, 3, and 6 months after completion of treatment

CONTACTS AND LOCATIONS:
Overall Officials: Michele Y Halyard, M.D., Study Chair — Mayo Clinic Mayo Clinic
Locations (1):
- Mayo Clinic in Arizona, Scottsdale, Arizona, United States